CLINICAL TRIAL: NCT03836625
Title: CareConekta: A Pilot Study of a Smartphone App to Improve Engagement in Postpartum HIV Care in South Africa
Brief Title: CareConekta: A Smartphone App to Improve Engagement in HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of Cape Town (Other); University of California, San Francisco (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate Clouse, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 181640; R34MH118028 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-02-11 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: HIV/AIDS; Pregnancy Related
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control arm will receive standard CareConekta, which will track their mobility with no additional features.
- Intervention (Experimental): The intervention arm will receive standard CareConekta, plus text notifications of nearby ART facilities when they have traveled >50 km from the study site for >7 days. At enrollment, participants in the intervention arm also will be able to opt-in to phone call(s) and/or WhatsApp message(s) from study staff to when they have met this travel threshold. The study staff calls and messages will ask about medication supply and will provide assistance with nearby facilities, if requested.
  Interventions: Other: CareConekta

INTERVENTIONS:
Other: CareConekta — CareConekta is a smartphone app that uses the phone's GPS to prospectively characterize mobility and allow for intervening in real-time. CareConekta uses the phone's built-in GPS system to record location coordinates.
  Arms: Intervention

SUMMARY:
Population mobility is common in South Africa, but important research gaps exist describing this mobility and its impact on engagement in HIV care, particularly among pregnant and postpartum women. Through this study, the investigators propose to test a smartphone application - CareConekta - to conduct essential formative work on mobility and evaluate this app as an intervention to facilitate engagement in HIV care during times of mobility. This work is critical to adapting CareConekta for widespread use, providing critical information about mobility during the peripartum period and the impact on engagement in HIV care, and piloting this intervention to improve engagement.

DETAILED DESCRIPTION:
South Africa is home to the world's largest antiretroviral therapy (ART) program, but sustaining high retention along the HIV care continuum has proven challenging in the country and throughout the wider region. Population mobility is common in South Africa, but important research gaps exist describing this mobility and its impact on engagement in HIV care. Postpartum women and their infants in South Africa are known to be at high risk of dropping out of HIV care after delivery and are frequently mobile. The investigators recently developed a beta version of a smartphone application (app) - CareConekta - that detects a user's smartphone location to allow for prospective characterization of mobility. Through this three-year study, the investigators propose to test CareConekta to conduct essential formative work on mobility and evaluate an intervention - the CareConekta app plus text notifications and optional staff phone calls and/or WhatsApp messages - to facilitate engagement in HIV care during times of mobility. After first adapting CareConekta to use appropriate smartphone technology for the local population, the investigators will characterize mobility among South African women during the peripartum period and its impact on engagement in HIV care. The investigators also will evaluate the acceptability, feasibility, and initial efficacy of using CareConekta as an intervention to improve engagement in HIV care. The investigators will work with a South African technology company with a strong connection to the South African Department of Health to adapt the app prior to enrolling study participants. The study will observe mobility within an observational cohort and will then assess the impact of the intervention among participants who travel during the study period. This work is critical to adapting an existing app for widespread use, providing critical information about mobility during the peripartum period and the impact on engagement in HIV care, and piloting an intervention to improve engagement. This study will lay the necessary groundwork for a larger efficacy trial of the intervention within different geographic settings.

ELIGIBILITY:
Inclusion Criteria:

1. We will only enroll participants attending the Gugulethu Community Health Centre, near Cape Town, South Africa
2. HIV-positive
3. adult (≥18 years)
4. pregnant (≥28 weeks)
5. own a smartphone that meets the technical requirements
6. willing to opt-in to installation of CareConekta on her personal phone and to mobility tracking
7. demonstrate the ability to read simple text language
8. willing to be randomized

Exclusion Criteria:

* If an interested participant meets all of the inclusion criteria, there are no additional exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We will enroll only pregnant women.
Enrollment: 200 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Clouse, PhD, MPH, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Gugulethu Community Health Centre, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be made available by request, subject to agreement to (1) a commitment to use the data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate computer technology and established security measures; (3) a plan for the dissemination of results; (4) appropriate authorship and recognition of all partners; and (5) a commitment to destroy or return the data after analyses are completed.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Anytime, by request

REFERENCES:
- [Derived] Noholoza S, Phillips TK, Madwayi S, Mrubata M, Camlin CS, Myer L, Clouse K. Smartphone Ownership and Usage Among Pregnant Women Living With HIV in South Africa: Secondary Analysis of CareConekta Trial Data. JMIR Form Res. 2023 Jun 22;7:e43855. doi: 10.2196/43855. PMID 37347521
- [Derived] Clouse K, Noholoza S, Madwayi S, Mrubata M, Camlin CS, Myer L, Phillips TK. The Implementation of a GPS-Based Location-Tracking Smartphone App in South Africa to Improve Engagement in HIV Care: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 May 19;11:e44945. doi: 10.2196/44945. PMID 37204838
- [Derived] Clouse K, Noholoza S, Ngcobo N, Madwayi S, Mrubata M, Camlin CS, Myer L, Phillips TK. Cohort profile: CareConekta: a pilot study of a smartphone application to improve engagement in postpartum HIV care in South Africa. BMJ Open. 2022 Nov 22;12(11):e064946. doi: 10.1136/bmjopen-2022-064946. PMID 36414286
- [Derived] Clouse K, Phillips TK, Camlin C, Noholoza S, Mogoba P, Naidoo J, Langford R, Weiss M, Seebregts CJ, Myer L. CareConekta: study protocol for a randomized controlled trial of a mobile health intervention to improve engagement in postpartum HIV care in South Africa. Trials. 2020 Mar 12;21(1):258. doi: 10.1186/s13063-020-4190-x. PMID 32164771

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 99 | 101
Completed | 84 | 89
Not Completed | 15 | 12
Not completed — Lost to Follow-up | 9 | 9
Not completed — Investigator withdrawn at/near time of enrollment | 6 | 1
Not completed — Death | 0 | 1
Not completed — Refused follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Total excludes 7 participants withdrawn by investigators at/soon after enrollment. Data were not included in analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 93 | 100 | 193
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 36] | 31 [28 to 35] | 32 [28 to 36]
Age, Customized [Count of Participants; unit: Participants]
  Age 18-24 years | 10 | 14 | 24
  Age 25-29 years | 22 | 21 | 43
  Age 30-34 years | 29 | 39 | 68
  Age 35 years and older | 32 | 26 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 100 | 193
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 93 | 100 | 193
Education [Count of Participants; unit: Participants]
  Never completed primary school | 1 | 1 | 2
  Primary school only | 5 | 3 | 8
  Some high school | 50 | 54 | 104
  Completed high school | 31 | 37 | 68
  Any tertiary education | 6 | 5 | 11
Employment [Count of Participants; unit: Participants]
  Currently employed | 34 | 42 | 76
  Not currently employed | 59 | 58 | 117
On antiretroviral therapy prior to first antenatal visit [Count of Participants; unit: Participants]
  No | 25 | 20 | 45
  Yes | 65 | 76 | 141
  Missing | 3 | 4 | 7
Birthplace [Count of Participants; unit: Participants]
  Western Cape Province, South Africa | 33 | 27 | 60
  In South Africa, but not Western Cape Province | 57 | 70 | 127
  Outside of South Africa | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mobility Prevalence
Description: The investigators will report the number of participants who travel during the study period (defined as 3 or more nights away from home), over the denominator of all participants who completed follow-up.
Time Frame: Baseline to End of Study (up to 2 years)
Population: The number of participants who reported travel during the study period (defined as 3 or more nights away from home)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Participants
  Traveled yes | 30 | 24
  Traveled no | 54 | 65

2. Primary Outcome: Median Number of Trips Per Person
Description: Among those who travel, the investigators will report the median and interquartile range number of trips during the study period.
Time Frame: Baseline to End of Study (up to 2 years)
Population: Participants who reported travel (n=54)
Measure: Median (Inter-Quartile Range); unit: trip
Arm/Group | Control | Intervention
Number analyzed (Participants) | 30 | 24
trip | 1 [1 to 1] | 1 [1 to 1]

3. Primary Outcome: CareConekta Feasibility: Same Phone at Follow-up
Description: The number of participants who report using the same phone from enrollment at follow-up
Time Frame: Baseline to End of Study (up to 2 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Participants
  No | 31 | 33
  Yes | 52 | 55
  Missing | 1 | 1

4. Secondary Outcome: Timing of Travel
Description: The investigators will determine timing of travel as it relates to delivery date, which will be obtained from participant questionnaire.
Time Frame: Baseline to End of Study (up to 2 years)
Population: Number of trips reported (n=60)
Measure: Count of Units; unit: Trips
Units Other Than Participants: Trips
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Number analyzed (Trips) | 33 | 27
Trips
  Traveled before delivery | 4 | 9
  Traveled after delivery | 29 | 18

5. Secondary Outcome: Permanent Move
Description: Was the move permanent (yes/no)
Time Frame: Baseline to End of Study (up to 2 years)
Population: Total number of trips per person, by study arm
Measure: Count of Units; unit: Trips
Units Other Than Participants: Trips
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Number analyzed (Trips) | 33 | 27
Trips
  Yes | 5 | 1
  No | 28 | 26

6. Secondary Outcome: CareConekta Feasibility: GPS Disabled During the Study Period
Description: The number of participants who disabled GPS during the study period
Time Frame: Baseline to End of Study (up to 2 years)
Population: The total number of participants who completed follow-up (n=173)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Participants
  No | 74 | 82
  Yes | 8 | 5
  I don't know | 1 | 1
  Missing | 1 | 1

7. Secondary Outcome: CareConekta Feasibility -- Participant Reported Sharing Phone
Description: The number of participants who reported sharing their phone with another person during the study period
Time Frame: Baseline to End of Study (up to 2 years)
Population: Total number of participants who completed follow-up (n=173)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Participants
  No | 77 | 71
  Yes | 7 | 18

8. Secondary Outcome: CareConekta Feasibility -- Participant Ever Opened App
Description: The number of participants who reported opening the CareConekta app at least once after enrollment visit
Time Frame: Baseline to End of Study (up to 2 years)
Population: All participants who completed follow-up (n=173)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
Participants
  No | 4 | 12
  Yes | 80 | 77

9. Secondary Outcome: CareConekta Feasibility -- Participant Used the App to Locate New Health Facilities
Description: The number of participants who reported using the CareConekta app to locate a new health facility.
Time Frame: Baseline to End of Study (up to 2 years)
Population: Number of participants who reported opening app during study period (n=157)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 80 | 77
Participants
  No | 69 | 68
  Yes | 11 | 9

10. Secondary Outcome: CareConekta Initial Efficacy -- Maternal Engagement in HIV Care
Description: The investigators will assess the initial efficacy of CareConekta as an intervention to improve engagement in HIV care. Efficacy will be assessed as the association (estimating adjusted hazard ratios) between study arm and maternal retention in care and viral suppression 6 months after delivery.
Time Frame: 6 months after delivery
Reporting Status: Not Posted

11. Secondary Outcome: CareConekta Initial Efficacy -- Infant Outcomes
Description: The investigators will assess the initial efficacy of CareConekta as an intervention to improve engagement in HIV care. Efficacy will be assessed as the association (estimating adjusted hazard ratios) between study arm and vertical HIV transmission and completion of 10-week infant HIV PCR test.
Time Frame: 10 weeks after delivery, study end
Reporting Status: Not Posted

12. Secondary Outcome: Impact of Mobility -- Maternal Engagement in HIV Care
Description: In the standard arm, the investigators will assess the association (estimating hazard ratios) between mobility during the study period and engagement in HIV care for the mother (defined as retention in care and viral suppression six months after delivery).
Time Frame: 6 months after delivery
Reporting Status: Not Posted

13. Secondary Outcome: Impact of Mobility -- Infant Outcomes
Description: In the standard arm, the investigators will assess the association (estimating hazard ratios) between mobility during the study period and completion of routine early infant diagnosis.
Time Frame: 10 weeks after delivery, study end
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout study period, median duration = 7.4 months
Description: Adverse events were reported per IRB and sponsor guidelines.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/93 | 1/100
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/100
Other Adverse Events (participants affected / at risk) | 0/93 | 0/100

LIMITATIONS AND CAVEATS:
We found that several key challenges impeded our study feasibility. The primary challenge is that during the study period, no participant's smartphone recorded at least one heartbeat per day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03836625/Prot_SAP_001.pdf